CLINICAL TRIAL: NCT00019383
Title: Immunization of Patients With Metastatic Melanoma Using Immunodominant Peptides From the Tyrosinase Protein or Tyrosinase Related Protein-1 (TRP1)
Brief Title: Vaccine Therapy in Treating Patients With Recurrent or Refractory Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065915; NCI-98-C-0022; NCI-T97-0088; NCT00001684 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-08-07 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2003-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant; sargramostim; tyrosinase-related protein-1

INTERVENTIONS:
Biological: aldesleukin
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Biological: tyrosinase peptide
Biological: tyrosinase-related protein-1

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Giving the vaccine with interleukin-2 or sargramostim may help kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of peptide vaccine with or without adjuvant interleukin-2 or sargramostim in treating patients who have recurrent or refractory metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether patients with refractory metastatic melanoma undergo partial or complete response to peptides specific to their HLA-antigen, either alone or when combined with 1 of 3 adjuvants.
* Evaluate the immunologic response to the peptide alone or when combined with 1 of 3 adjuvants in these patients.

OUTLINE: Patients are stratified by HLA status (A1 vs A3 vs A24 vs A31).

Patients are assigned to 1 of 4 vaccine groups:

* Group 1 (HLA-A1 positive): Patients receive tyrosinase:240-251.
* Group 2 (HLA-A3 positive): Patients receive gp100:17-25. (closed to accrual 5/17/2000)
* Group 3 (HLA-A24 positive): Patients receive tyrosinase:206-214.
* Group 4 (HLA-A31 positive): Patients receive tyrosinase related protein-1. Each peptide vaccine is separately emulsified in Montanide ISA-51 and administered subcutaneously into the thigh. Patients are treated with peptide vaccine alone or combined with 1 of 3 possible adjuvants (interleukin-2 (IL-2) IV, IL-2 delayed IV, or sargramostim (GM-CSF) SQ) depending on the time of entry into study and response to treatment.

At least 4 to 6 patients are accrued for the peptide alone cohort before beginning accrual on the other cohorts. Any patient who experiences unacceptable toxicity due to adjuvant therapy is taken off study. If a second patient develops unacceptable toxicity, that schedule of peptide administration is discontinued.

Patients exhibiting stable, minor, mixed, or partial response may receive up to 12 additional courses.

Patients are followed for 4-6 weeks.

PROJECTED ACCRUAL: A maximum of 457 patients will be accrued for this study over 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven refractory metastatic melanoma

  * Must be HLA-A1, HLA-A3, HLA-A24, or HLA-A31 positive
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance Status:

* ECOG 0-1

Life Expectancy:

* Greater than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3
* No coagulation disorder

Hepatic:

* AST or ALT less than 2 times upper limit of normal
* Bilirubin no greater than 1.6 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No major cardiovascular disease

Pulmonary:

* No major respiratory disease

Other:

* Not pregnant
* Fertile patients must use effective contraception
* HIV negative
* Hepatitis B surface antigen negative
* No known allergy to Montanide ISA-51
* No active systemic infection
* No immunodeficiency disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy
* No concurrent biologic therapy

Chemotherapy:

* At least 3 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy
* No concurrent steroid therapy or other endocrine therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Prior or concurrent surgery for melanoma allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States